CLINICAL TRIAL: NCT02376972
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of Rifaximin Vaginal Tablets in the Treatment of Bacterial Vaginosis
Brief Title: Efficacy and Safety Study of Rifaximin Vaginal Tablets in Bacterial Vaginosis
Acronym: VARIANT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: According to the Recommendation of the Indipendent Data Monitoring Committee
Sponsor: Alfasigma S.p.A. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RFX-VAG/003/2012
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: BACTERIAL VAGINOSIS
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Benchmarking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RIFAXIMIN VAGINAL TABLET 25 MG (Experimental): RIFAXIMIN VAGINAL TABLET 25 MG ADMINISTERED ONCE A DAY FOR 5 DAYS
  Interventions: Drug: RIFAXIMIN VAGINAL TABLET 25 MG
- RIFAXIMIN VAGINAL TABLET 100 MG (Experimental): RIFAXIMIN VAGINAL TABLET 100 MG ADMINISTERED ONCE A DAY FOR 5 DAYS
  Interventions: Drug: RIFAXIMIN VAGINAL TABLET 100 MG
- PLACEBO VAGINAL TABLET (Placebo Comparator): PLACEBO VAGINAL TABLET ADMINISTERED ONCE A DAY FOR 5 DAYS
  Interventions: Drug: PLACEBO VAGINAL TABLET
- METROGEL VAGINAL (Active Comparator): METROGEL VAGINAL ADMINISTERED ONCE A DAY FOR 5 DAYS
  Interventions: Drug: METROGEL VAGINAL

INTERVENTIONS:
Drug: RIFAXIMIN VAGINAL TABLET 25 MG — RIFAXIMIN VAGINAL TABLET 25 MG O.D./5 DAYS INTRAVAGINALLY
  Arms: RIFAXIMIN VAGINAL TABLET 25 MG
Drug: RIFAXIMIN VAGINAL TABLET 100 MG — RIFAXIMIN VAGINAL TABLET 100 MG O.D./5 DAYS INTRAVAGINALLY
  Arms: RIFAXIMIN VAGINAL TABLET 100 MG
Drug: PLACEBO VAGINAL TABLET — PLACEBO VAGINAL TABLET O.D./5 DAYS INTRAVAGINALLY
  Arms: PLACEBO VAGINAL TABLET
Drug: METROGEL VAGINAL — METROGEL VAGINAL O.D./5 DAYS INTRAVAGINALLY
  Arms: METROGEL VAGINAL

SUMMARY:
THE STUDY HAS BEEN DESIGNED TO COMPARE THE EFFICACY OF TWO DOSES (25 MG AND 100 MG) OF RIFAXIMIN VAGINAL TABLETS VERSUS PLACEBO IN SUBJECTS WITH BACTERIAL VAGINOSIS

DETAILED DESCRIPTION:
THIS IS A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED STUDY PLANNING TO ENROL 626 SUBJECTS AFFECTED BY BACTERIAL VAGINOSIS.

PRIMARY ENDPOINT:

TO COMPARE THE EFFICACY OF TWO DOSES (25 MG AND 100 MG) OF RIFAXIMIN VAGINAL TABLETS VERSUS PLACEBO IN SUBJECTS WITH BACTERIAL VAGINOSIS

SECONDARY ENDPOINT:

TO COMPARE THE EFFICACY OF TWO DOSES (25 MG AND 100 MG) OF RIFAXIMIN VAGINAL TABLETS VERSUS METROGEL VAGINAL IN SUBJECTS WITH BACTERIAL VAGINOSIS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bacterial vaginosis with Amsel's criteria (4 out of 4 fulfilled criteria):

  * Off white (milky or gray), thin, homogeneous, adherent vaginal discharge
  * pH >4.5
  * Positive "whiff test"
  * Presence of clue cells ≥20%
* Bacteriological diagnosis of bacterial vaginosis with Gram stain Nugent score ≥ 4 (patients may be enrolled/randomized without this result)
* Post-menarchal, pre-menopausal female patient
* Non-pregnant (negative urine pregnancy test at Entry Visit/V1) nor breast-feeding patient
* Patient aged between 18 50 years, inclusively
* Patient who is willing to be asked questions about personal medical health and sexual history
* Patient capable of and willing to conform to the study protocol
* Patient who have been thoroughly informed of the aim of the study and the study procedures and who provided signed and dated written informed consent form
* Patient who agrees to abstain from intercourse during the 5 day treatment period
* Patient who agrees also to abstain from intercourse 3 days before the scheduled visits of follow-up
* Patient who agrees to abstain from the use of any other intravaginal product (i.e., douching, feminine deodorants sprays, tampons, spermicides, gels, foams, vaginal birth control ring and diaphragms) during the entire study period
* Patient who agrees to use an adequate method of birth control for the duration of the study to avoid pregnancy. Acceptable methods include a history of bilateral tubal ligation, male partner with a vasectomy, a hormonal contraceptive [oral, patch, injectable or implantable (excluding intrauterine implantable devices [IUD], intrauterine system [IUS] and vaginal rings), or abstinence
* Patient who agrees to abstain from alcohol ingestion during the 5-day treatment period and for 1 day afterward

Exclusion Criteria:

* Virginity
* Patient with other infectious causes of vulvovaginitis (e.g., candidiasis, Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae, active Herpes simplex lesions, or Human Papilloma Virus lesions); patients may be enrolled/randomized without these results)
* Other vulvovaginal or cervical conditions, abnormalities or disorders confounding the interpretation of clinical response (including total hysterectomy)
* Symptoms suggestive of pelvic inflammatory disease
* Patient with intra uterine device (IUD), intrauterine system (IUS), or vaginal ring as contraceptive method
* Patient with severe hepatic insufficiency (Child C)
* Patient with severe cardiac insufficiency (NYHA - New York Heart Association classes 3 - 4)
* Patient who will be being evaluated, including colposcopy and cervical biopsies, or being treated during the study period, for abnormal Pap test or cervical carcinoma. To note that if the Pap test will be performed at baseline, the result will be known after the randomization visit: patients may be enrolled without this result
* Any condition or circumstance that would prevent completion of the study or interfere with analysis of study results, including a history of drug or alcohol abuse, mental illness or non-compliance with treatments or visits, immunological (including HIV infection), hematological or neoplastic disease (including all cervical neoplastic diseases)
* Cervical cryotherapy, loop electrosurgical excision (LEEP), cervical laser, or any other ablative or excisional cervical procedures within the last 3 months
* Vaginal laser within the last 3 months
* Patient with clinically relevant pathological laboratory values
* Known hypersensitivity to rifaximin
* Known hypersensitivity to excipients present in rifaximin, placebo or metronidazole formulations
* Known hypersensitivity to metronidazole, either orally or topically administered, or any forms of parabens
* Concurrent anticoagulant therapy with coumadin or warfarin
* Menstruating or anticipated menstruation/withdrawal bleed at Entry Visit/V1 and during the drug administration
* Patient who received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days of randomization
* Patient who have participated in another clinical trial or have taken an investigational drug within the last 4 weeks prior screening
* Patient who has taken disulfuram within the last 14 days
* Withdrawal of informed consent
* Patient previously randomized in this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 392 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
CLINICAL CURE OF BACTERIAL VAGINOSIS | Day 22-30
  RESOLUTION OF 3 OUT OF 4 AMSEL'S CRITERIA, I.E. NORMAL PHYSIOLOGICAL DISCHARGE, NEGATIVE "WHIFF TEST", CLUE CELLS >20%

SECONDARY OUTCOMES:
BACTERIOLOGICAL CURE OF BACTERIAL VAGINOSIS | Day 22-30
  GRAM STAIN NUGENT SCORE <4
THERAPEUTIC CURE OF BACTERIAL VAGINOSIS | Day 22-30
  AMSEL'S CRITERIA AND GRAM STAIN NUGENT (RESOLUTION OF 3 OUT OF 4 AMSEL'S CRITERIA AND NUGENT SCORE <4)
MAINTENANCE OF CLINICAL CURE OF BACTERIAL VAGINOSIS | Day 61-70
  AMSEL'S CRITERIA (RESOLUTION OF 3 OUT OF 4 AMSEL'S CRITERIA)
MAINTENANCE OF BACTERIOLOGICAL CURE OF BACTERIAL VAGINOSIS | Day 61-70
  NUGENT SCORE <4
MAINTENANCE OF THERAPEUTIC CURE OF BACTERIAL VAGINOSIS | 60-69 DAYS AFTER THE FIRST DAY OF TREATMENT
  AMSEL'S CRITERIA AND NUGENT SCORE (MAINTENANCE OF RESOLUTION OF 3 OUT OF 4 AMSEL'S CRITERIA AND NUGENT SCORE <4)
NUMBER, INTENSITY AND TYPE OF ADVERSE EVENTS | Up to Day 70
  The incidence of adverse events to be summarized by body system and MedDRA preferred term.
LOCAL OBJECTIVE TOLERABILITY | Day 22-30
  Vaginal mucosa status in terms of erythema (score 0 to 3), edema (score 0 to 3), pethechial hemorrhages (absence/presence), ulcers (absence/presence)
LOCAL SUBJECTIVE TOLERABILITY | Day 1 to Day 5
  Grade (from 0 to 4) of vaginal itching, pain and burning

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Tacchi, MD, Study Director — Alfasigma S.p.A.
Locations (1):
- College of Medicine Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided